CLINICAL TRIAL: NCT03840655
Title: Fluorescent Thoracoscopy Used in Surgery for Palmar Hyperhidrosis
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Jun Wang, Department Chief, Peking University People's Hospital
Other Study IDs: 2017PHB101-01
Record Dates: First submitted 2019-02-09; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Palmar Hyperhidrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- palmar hyperhidrosis: VATS R4 Sympathicotomy performed on all patients. Fluorescent thoracoscopy was used to identify the shifting mode of sympathetic ganglions.
  Interventions: Procedure: Near-Infrared Imaging Thoracoscopy

INTERVENTIONS:
Procedure: Near-Infrared Imaging Thoracoscopy — Sympathicotomy performed by near-infrared imaging thoracoscopy

SUMMARY:
T3/T4 endoscopic thoracic sympathicotomy is a widely accepted and effective treatment for primary palmar hyperhidrosis. However, sympathetic ganglions are invisible with traditional thoracoscopy and until now, the location of ganglions are confirmed by rib indirectly. The team from thoracic department of Peking University People's Hospital discovered that the sympathetic ganglions can be visualized with fluorescent thoracoscopy. Thus, investigators want to apply fluorescent thoracoscopy in sympathicotomy of palmar hyperhidrosis, to conduct a more precise operation and compare the efficiency of the novel and traditional methods.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with primary palmar hyperhydrosis.
2. Accept surgical treatment and signed informed consent.

Exclusion Criteria:

1. Liver dysfunction.
2. Allergic to indocyanine green.
3. Can't tolerate thoracoscopic surgery.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients suffering from primary palmar hyperhidrosis
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Anatomical variation of the sympathetic ganglions | during surgery
  Record the spatial relationship between sympathetic ganglions and ribs, for example: T3/R4 represents the T3 sympathetic ganglion is located on the 4th rib.

SECONDARY OUTCOMES:
Improvement of palmar sweating | 1 month after surgery
  Use questionnaire including 3 descriptive names of scale ( over dry, comfortable and wet) to record the surgical effect on palmar sweating.
Degree of compensatory hyperhidrosis | 1 month after surgery
  Use questionnaire including 4 descriptive names of scale ( none, mild, moderate and severe) to record the side effect (compensatory hyperhidrosis) of this surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People'S Hospital, Beijing, Beijing Municipality, China